CLINICAL TRIAL: NCT07233031
Title: ROLE OF DESIGNED PROGRAM IN UNIVERSAL EXERCISE UNIT ON UPPER LIMB IN CHILDREN WITH SPASTIC HEMIPLEGIA
Brief Title: Effectiveness of Universal Exercise Unit Exercise on Upper Limb Strength Using Biodex Isokinetic
Acronym: UEU/CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samaa Hussein Rajab, assistant lecturer in physical therapy faculty, department of pediatric and its surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004849
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy Spastic Hemiplegic
Keywords: universal exercise unit , muscle strength

STUDY DESIGN:
Intervention Model Description: for group A: The session time ranged between 50-60 minutes according to child cooperation and numbers of repetitions the child could do for group B: Each child performed 1 or 2 sets of 8-15 repetitions with a light to moderate load (about 60% 1- RM)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (standard treatment) (Active Comparator): children in control group received standard physiotherapy
  Interventions: Other: Control (Standard treatment)
- experimental (Experimental): a designed physical therapy program in Universal exercise that began with testing one repetition maximum (1-RM). One repetition maximum (1-RM) was determined through the chest press. children had been targeted upper limb strengthening program
  Interventions: Procedure: Experimental

INTERVENTIONS:
Procedure: Experimental — designed physical therapy program in Universal exercise unit for strengthening upper limb. fundamental beginning position for every exercise. Total session time in the UEU was approximately 30 minutes.
  The resisted exercise targeted shoulder flexor and extensor muscles, shoulder abductor and adductor muscles and for elbow extensor muscles
  Arms: experimental
Other: Control (Standard treatment) — traditional physio therapy program.
  Arms: control (standard treatment)

SUMMARY:
The aim of the study is to determine the role of designed program in the universal exercise unit on upper limb function and strength in children with spastic hemiplegia. forty children with spastic hemiplegia cerebral palsy from both sexes had been selected from the Outpatient Clinic of the Faculty of Physical Therapy, Cairo University . Children were divided into two groups of equal numbers; 20 patients in each group. Group A: Children in this group received a selected physical therapy program. Group B: Children in this group received a designed physical therapy program in UEU in addition to the selected physical therapy program. A-Materials for evaluation 1- For the Quality Of Upper Extremity Skill Test (QUEST),2- Biodex Isokinetic systems.Evaluation was carried out for each child individually before and after 3 months of treatment

DETAILED DESCRIPTION:
This study is designed to answer the following question:

Is there an effect of designed program in universal exercise unit on upper limb function and strength in children with spastic hemiplegia? Purpose of The Study The purpose of the study is to determine the role of designed program in the universal exercise unit on upper limb function and strength in children with spastic hemiplegia.

Null Hypothesis Is there is no role of designed program in the universal exercise unit on the upper limb in children with spastic hemiplegia.

The study was concluded forty children with spastic hemiplegic cerebral palsy from both sexes had been selected from according to the following criteria:

* children ages were ranged from 5-9 years old.
* The children had spasticity grades 1, 1+ degree according to Modified Ashworth scale
* The children were selected to be in level I and II GMFCs
* The children were selected to be in level II MACs participants had been excluded if they had the following:

  1. Visual or hearing impairment
  2. Orthopedic surgery of upper limbs for the last 6 months
  3. Cardiopulmonary diseases Children were equally assigned into two groups using simple randomization, control group (A) and study group (B). Each group would consist of 20 children with spastic hemiplegia CP.

Group (A): Children in this group received a selected physical therapy program. Group (B): Children in this group received the selected physical therapy program in addition to a designed physical therapy program in UEU.

Evaluation was carried out for each child individually before and after 3 months of treatment.

A-For Assessment

1. The Quality of Upper Extremity Skill Test (Quest) The QUEST test included 34 items in four domains of (dissociated movement, grasp, weight bearing and protective extension).

   Each child was instructed to hold the position for at least two seconds. The total testing timing including the administration and scoring was approximately 45 minutes.

   The scoring was performed and recorded in scoring box. Even if the item was not tested (I.e: yes, no, not tested)
2. The Biodex Isokinetic system The testing session had been started with a warm up procedure, consisting of shoulder movements in all directions, push up-exercises against the wall and stretching. For the testing procedure, the closed chain attachment was fixed to the isokinetic dynamometer in a horizontal position. Essentially, this device converts rotational motion at the dynamometer into linear motion, allowing closed kinematic chain or linear movements The evaluation was carried out for each child individually before and after three month of treatment.

Tested muscles were elbow flexors, elbow extensor, shoulder flexors, shoulder extensors.

ELIGIBILITY:
Inclusion Criteria:

* Their ages were ranged from 5-9 years old.
* They had spasticity grades 1, 1+ degree according to Modified Ashworth scale
* They were selected to be in level I and II GMFCs They were selected to be in level II MACs

Exclusion Criteria:

* Visual or hearing impairment
* Orthopedic surgery of upper limbs for the last 6 months
* Cardiopulmonary diseases

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
The Quality of Upper Extremity Skill Test | The total testing timing including the administration and scoring was approximately 45 minutes. The scoring was performed and recorded in scoring box. Even if the item was not tested (I.e: yes, no, not tested)
  The Quality of Upper Extremity Skill est test included 34 items in four domains of dissociated movement, grasp, weight bearing and protective extension. All children in this study were assessed in the four domains. The total number of 'yes' and 'no' responses provide the raw score for each domain. This is then weighted and transformed into a final score range of zero to 100.

SECONDARY OUTCOMES:
The Biodex Isokinetic system | The evaluation was carried out for each child individually before and after three month of treatment.
  The testing session had been started with a warm up procedure, consisting of shoulder movements in all directions, push up-exercises against the wall and stretching Tested muscles were elbow flexors, elbow extensor, shoulder abductors, shoulder adductors

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa A Zaky, professor, Study Director — Cairo University
Locations (1):
- Outpatient Clinic of the Faculty of Physical Therapy, Cairo University's, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No